CLINICAL TRIAL: NCT04612530
Title: Irreversible Electroporation and Nivolumab Combined With Intratumoral Administration of a Toll-like Receptor Ligand as a Means of in Vivo Vaccination for Oligometastatic Pancreatic Ductal Adenocarcinoma
Brief Title: PANFIRE-3 Trial: Assessing Safety and Efficacy of Irreversible Electroporation (IRE) + Nivolumab + CpG for Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Dr. M.R. Meijerink, Professor of Interventional Oncology, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.231 - NL73415.029.20
Record Dates: First submitted 2020-09-09; First posted 2020-11-03 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Pancreatic Cancer; Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; metastatic pancreatic cancer; pancreatic ductal adenocarcinoma; metastatic pancreatic ductal adenocarcinoma; PDAC
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation; Nivolumab; Toll-Like Receptor 9

STUDY DESIGN:
Intervention Model Description: Step-up design. Arms A (monotherapy Nivolumab, 6 patients) and B (IRE + Nivolumab, 6 patients) will open first. A safety and toxicity analysis will be performed after the inclusion of patient 6 and patient 12. Arm C (CpG + IRE + Nivolumab, 6 patients) will open if the interim results demonstrate safety of arms A and B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: Nivolumab (Active Comparator): 4 weeks after pre-treatment with FOLFIRINOX (4-8 cycles), the patient will start with the Nivolumab scheme. The first month, a biweekly dose of 240 mg will be administered, followed by a monthly dose of 480 mg. This treatment will continue until disease progression.
  Interventions: Drug: Nivolumab
- Arm B: IRE + Nivolumab (Experimental): 4 weeks after pre-treatment with FOLFIRINOX (4-8 cycles), the patient will first receive (an incomplete) IRE of the primary pancreatic tumor. 2 weeks thereafter, they will start the Nivolumab scheme. The first month, a biweekly dose of 240 mg will be administered, followed by a monthly dose of 480 mg. This treatment will continue until disease progression.
  Interventions: Device: Irreversible Electroporation (IRE); Drug: Nivolumab
- Arm C: CpG + IRE + Nivolumab (Experimental): 4 weeks after pre-treatment with FOLFIRINOX (4-8 cycles), a toll-like receptor ligand (CpG) will be administered into the primary pancreatic tumor. A week later, the patient will receive (an incomplete) IRE of the primary tumor. 2 weeks thereafter, they will start the Nivolumab scheme. The first month, a biweekly dose of 240 mg will be administered, followed by a monthly dose of 480 mg. This treatment will continue until disease progression.
  Interventions: Device: Irreversible Electroporation (IRE); Drug: Nivolumab; Drug: Toll-Like Receptor 9

INTERVENTIONS:
Device: Irreversible Electroporation (IRE) — Irreversible electroporation (IRE) is a local ablative technique that utilizes electrical pulses to destroy tumor tissue
  Arms: Arm B: IRE + Nivolumab; Arm C: CpG + IRE + Nivolumab
Drug: Nivolumab — Nivolumab is an immune checkpoint inhibitor targeting the PD-1 receptor on T-cells. Binding of the PD-1 monoclonal antibody onto the PD-1 receptor blocks the brake signal on the T-cells, allowing them to attack the cancer cells.
Drug: Toll-Like Receptor 9 — Toll-Like Receptor 9 (CpG) is an oligodeoxynucleotide that stimulates dendritic cells to release IFN type I, activating natural killer and infiltrating T cells. This creates a more pro-immunogenic tumor environment.
  Arms: Arm C: CpG + IRE + Nivolumab

SUMMARY:
Irreversible electroporation is a local ablative technique used in the treatment of pancreatic cancer. In addition to its cytoreductive ability, IRE also induces a systemic immune response. However, this immune response is not potent enough to establish durable regression of the tumor. The immune response can be leveraged by combining IRE with immunotherapy. The primary aim of this study is to determine the safety of IRE + Nivolumab (arm B) and IRE + Nivolumab + CpG (arm C). The secondary aim is to assess efficacy of the experimental arms (B, C) and control arm A (Nivolumab monotherapy), based on overall and progression-free survival as well as locoregional and systemic immune modulation.

DETAILED DESCRIPTION:
Pancreatic carcinoma is one of the deadliest types of cancer. In contrast to other cancers, new treatment options have demonstrated only moderate improvements for pancreatic cancer in terms of overall survival. Patients with metastasized disease (stage IV, AJCC) that are treated with chemotherapy in the Netherlands currently present a median overall survival of 6.4 months. Previous research has shown promising results for patients with locally advanced pancreatic cancer (LAPC, stage III, AJCC) with regards to combination treatment with chemotherapy and irreversible electroporation (IRE), a local ablation technique that utilizes electrical pulses to destroy cancerous tissue. In addition to an increase in overall survival, IRE induced a systemic immune response. However, the immune response was not potent enough to generate a lasting anti-tumor effect. Leveraging the body's own immune response by using local and systemic immunotherapy may create a synergistic effect, potentially inducing a durable anti-tumor response. The PANFIRE-III is a prospective randomised phase 1 trial with the primary aim to determine safety of the combination therapies IRE + Nivolumab (arm B) and CpG + IRE + Nivolumab (arm C) in patients with oligo-metastasized pancreatic cancer. The secondary goal is to determine efficacy of the experimental arms (arm B, C) compared to the control arm A (Nivolumab monotherapy). This will be assessed by looking at the overall and progression-free survival as well as the locoregional and systemic immune response. The treatment combination of IRE with immunotherapy has the potential to generate systemic protection by in vivo vaccination against pancreatic cancer cells, hereby inhibiting both local and distant tumor growth.

ELIGIBILITY:
Inclusion Criteria:

* Radiological and histopathologically proven stage IV pancreatic cancer (according to the AJCC staging system for pancreatic cancer);
* Primary oligometastatic disease, defined as at least 1 hepatic metastasis but occurrence of other metastases is not necessarily restricted to the liver, maximum of metastases is to be determined on a case by case basis by the multidisciplinary tumor board.
* Primary tumor is in situ.
* A minimum of 4 cycles of FOLFIRINOX chemotherapy is required but with the explicit aim to strive for completion of 8 cycles of FOLFIRINOX before study inclusion, with at least stable disease on CTscan.
* Age ≥ 18 years.
* World Health Organisation scale (WHO) performance status 0 - 2;
* Adequate bile drainage in case of biliary obstruction.

Exclusion Criteria:

* Trans-mucosal tumor invasion into surrounding duodenum or stomach;
* Active epilepsy (last convulsion < 5 years);
* History of cardiac disease:

  * Congestive heart failure > NYHA Class 2
  * Active coronary artery disease (defined as myocardial infarction within 6 months prior to screening);
  * Ventricular cardiac arrhythmias requiring anti-arrhythmic therapy or pacemaker (beta blockers for antihypertensive regimen are permitted; atrial fibrillation is not contra-indicated);
* Known hypersensitivity to any oligodeoxynucleotides.
* Compromised liver function defined as warning signs of portal hypertension, INR > 1,5 without use of anticoagulants, bilirubin > x 1.5 Upper limit of normal range (ULN) ASAT >3.0 x ULN, ALAT >3.0 x ULN.
* Compromised kidney function defined as eGFR <30 ml/min (using the Cockcroft Gault formula);
* Active autoimmune disease requiring disease-modifying therapy at the time of screening: i.e. > 10 mg prednisolone per day or equivalent to this regimen.
* Uncontrolled hypertension. Blood pressure must be ≤160/95 mmHg at the time of screening on a stable antihypertensive regimen;
* Uncontrolled infections (> grade 2 NCI-CTC version 3.0); requiring antibiotics
* Pregnant or breast-feeding subjects; Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment;
* Immunotherapy prior to the procedure for the treatment of cancer;
* Previous surgical therapy for pancreatic cancer;
* Second primary malignancy with median 5 year OS < 90%, this excludes adequately treated cancers like: non-melanoma skin cancer, in situ carcinoma of the cervix uteri, superficial bladder cancer or other malignancies treated previously without signs of recurrence.
* Allergy to contrast agent.
* Allergy to PET tracers 18F-FDG and 18F-BMS-986192 Zr-89-Nivolumab
* Any implanted stimulation device;
* Portal vein or VMS stenosis > 70% (relative contra-indication)
* Any condition that is unstable or that could jeopardize the safety of the subject and their compliance in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the combination treatment IRE + immunotherapy based on adverse events | From randomization until 1 year later
  Determined by the treatment related (serious) adverse events

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until death, assessed up to 5 years
  Overall survival in terms of months
Progression-Free Survival | From date of randomization until unequivocal disease progression, assessed up to 5 years
  Progression-free survival in terms of months
Immunomodulation (local) | Biopsies taken at T=0 (prior to treatment), T=2 weeks and T=6 weeks
  The local immune response will be assessed using flow cytometry and immunohistochemistry of 2 biopsies (1x primary, 1x metastasis). Markers include those of T-cells, dendritic cells and others.
Immunomodulation (systemic) | Blood taken at T=0 (prior to treatment), T=2 weeks and T=6 weeks
  The systemic immune response will be assessed using flow cytometry of peripheral blood. Markers include those of T-cells, dendritic cells, MDSCs, NK cells.
Tumor Response on Imaging | PET scans at T= 0 (prior to treatment), T= 6 weeks and T=3months. CT scans will be made at T= 0 (prior to treatment), T= 6 weeks, T=3months, followed by a scan every subsequent 3 months (T=6m,9m,12m etc) until unequivocal disease progression.
  Tumor response will be assessed using PET-CT scans: tracer uptake of FDG and PD-L1. CT scans will be employed to determine tumor response based on the RECIST criteria.
Quality of Life throughout treatment based on overall health | Quality of Life will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  Based on the following EORTC questionnaire: EQ-5D-L5. Question types include: scale 1-5
Quality of Life throughout treatment based on specific health questions | Quality of Life will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  Based on the following EORTC questionnaire: QLQ-C30 Question types include: scale 1-5, scale 1-7
Quality of Life throughout treatment based on Chemotherapy-Induced Peripheral Neuropathy | Quality of Life will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  Based on the following EORTC questionnaire: QLQ-CIPN20 Question types include: scale 1-4
Quality of Life throughout treatment specifically in patients with pancreatic cancer | Quality of Life will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  Based on the following EORTC questionnaire: QLQ-PAN26 Question types include: scale 1-4
Quality of Life throughout treatment based on the patient's happiness and emotional functioning | Quality of Life will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  Based on the following questionnaire: QLQ-HAPINES Question types include: scale 1-10
Quality of Life throughout treatment based on anxiety and depression | Quality of Life will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  Based on the following questionnaire: QLQ-HADS Question types include: scale 1-4
Quality of Life throughout treatment based on a patient's psychological state regarding their disease | Quality of Life will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  Based on the following questionnaire: QLQ-WOPS Question types include: scale 1-4, scale 1-10, yes/no, open
Quality of Life throughout treatment based on (decreased) pancreatic functionality | Quality of Life will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  Based on the following questionnaire: EPI Question types include: 5 optional answers, scale, 1-4, scale 1-5, yes/no, open
Pain based on the Visual Analog Score (VAS) | Pain will be assessed every 3 months (T=0 (baseline), T=3months, etc) up to 1 year
  The pain questionnaire is based on the VAS and includes scale type questions (1 - 10) with higher scores referring to more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn R Meijerink, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam University Medical Centre (location VUmc), Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No